CLINICAL TRIAL: NCT02816749
Title: Maggot Debridement Therapy Versus Conventional Dressing Therapy to Treat Type 2 Diabetic Mellitus Foot Ulcers: A Prospective Randomized Controlled Study
Brief Title: Maggot Debridement Therapy Versus Conventional Dressing Therapy to Treat Diabetic Foot Ulcers
Acronym: MDTDF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DMUF-01
Record Dates: First submitted 2016-04-26; First posted 2016-06-29 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetic Foot; Wound Healing; Larva; Occlusive Dressings
MeSH Terms: conditions — Diabetic Foot | interventions — Maggot Debridement Therapy; Occlusive Dressings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maggot debridement therapy(MDT) (Experimental): Participant will receive bio-bags treatment every 3 days until the wound heal completely, when wounds assessed.
  Interventions: Procedure: Maggot debridement therapy
- Conventional Dressing Therapy(CDT) (Active Comparator): Participant will be disinfected by iodophor and dressed by gauze 3 days until the wound heal completely, when wounds assessed.
  Interventions: Procedure: Conventional Dressing Therapy

INTERVENTIONS:
Procedure: Maggot debridement therapy — Participant will receive bio-bags treatment every 3 days until the wound heal completely, when wounds assessed.
  Other Names: MDT; Maggot Therapy; Larvae Therapy
  Arms: Maggot debridement therapy(MDT)
Procedure: Conventional Dressing Therapy — Participant will be disinfected by iodophor and dressed by gauze 3 days until the wound heal completely, when wounds assessed.
  Other Names: CDT; Occlusive Dressings; Dressing Therapy
  Arms: Conventional Dressing Therapy(CDT)

SUMMARY:
This is a prospective study of participants with diabetic foot ulcers who will receive either maggot debridement therapy (MDT) or conventional dressing therapy (CDT). Wound healing time is the main outcome measure to compare the clinical efficacy of these two therapies. The investigators developed a hypothesis that MDT could achieve remarkable shorter time and better healing rate for wound closure when compared with CDT.

DETAILED DESCRIPTION:
The investigators designed a prospective randomized study to compare the clinical safety and efficacy of maggot debridement therapy (MDT) and conventional dressing therapy (CDT). This study is scheduled from July 2016 to February 2017. Patients, aged from 18-80, who suffered from type 2 diabetic mellitus foot ulcers with Grade 1 or Grade 2 according to the Wagner classification could be the participants of this study. A sample of 138 participants was calculated based on the morbidity of diabetic foot ulcers, accounting for estimated 10% attrition rate. The glycemic control is important for the validity of study results. A specific team of endocrine doctors will manage the blood glucose of participants of two groups within the range of 7-10 mmol/L.

Participants will be allocated into MDT group and CDT group randomly according to the random number table. For MDT-participants, bio-bags containing sterilized, live, medicinal Lucilia sericata larvae will be placed on the wound of ulcers. For CDT-participants, conventional dressing (disinfected by iodophor, dressed by gauze ) will be performed ordinally. Every 3 days the procedures of two groups will be performed and wounds assessment will be done until the wounds closure is achieved. The wounds assessment, including measurement of the area of wound surface and bacterial culture, will be performed by a specific team of microsurgical doctors. The outcome measures include wound healing time (days) and the time negative bacterial culture occurs (days). The secondary outcome measures include the area of wound surface (cm2), treatment related pain, comfort of the dressing and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged from 18-80 years old.
2. Participants with type 2 diabetes mellitus longer than one year, foot ulcer longer than three weeks and with ischemic symptoms of lower limb.
3. The ulcer erosion depth is not reached and muscle layer.
4. The Wagner classification of ulcers should be Grade 1 or Grade 2.
5. Blood glucose control: Fasting blood glucose ≤ 8mmol / L; Postprandial blood glucose two hours ≤ 11.1 mmol / L.
6. Participants do not receive ulcer wound management in the past three days when recruited.
7. Participants with neuropathy symptoms, such as limb numbness, tingling or pain, especially pain at night.

Exclusion Criteria:

1. Participants with acute thrombosis that required thrombolysis or thrombectomy.
2. Participants with severe systemic infection.
3. Participants who are sensitive to pain.
4. Participants with bone/joint deformities of foot (eagle claw toes, hammer toes)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Wound healing time(days) | From date of randomization until the date of the complete closure of wound or up to 12 weeks, whichever came first.
  Wound complete closure is achieved.

SECONDARY OUTCOMES:
Area of wounds (cm2) | From date of randomization until the date of the complete closure of wound or up to 12 weeks, whichever came first.
  Area of wounds are measured by transparency-based digital imaging method.Every 3/4 days when procedures(bio-bags/dressings) given.
Adverse events | From date of randomization until the date of the complete closure of wound or up to 12 weeks, whichever came first.
  Adverse events such as allergic reaction, infection, local pain and escape of the larvae from bio-bag.Every 3/4 day when procedures(bio-bags/dressings) given.
Negative bacterial culture time (days) | From date of randomization until the date of the complete closure of wound or up to 12 weeks, whichever came first.
  The time that negative bacterial culture occured from recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Shou-Yu Wang, Dr, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (2):
- China (2):
  - the Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - the First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pinheiro MA, Ferraz JB, Junior MA, Moura AD, da Costa ME, Costa FJ, Neto VF, Neto RM, Gama RA. Use of maggot therapy for treating a diabetic foot ulcer colonized by multidrug resistant bacteria in Brazil. Indian J Med Res. 2015 Mar;141(3):340-2. doi: 10.4103/0971-5916.156628. PMID 25963495
- [Background] Sun X, Jiang K, Chen J, Wu L, Lu H, Wang A, Wang J. A systematic review of maggot debridement therapy for chronically infected wounds and ulcers. Int J Infect Dis. 2014 Aug;25:32-7. doi: 10.1016/j.ijid.2014.03.1397. Epub 2014 May 16. PMID 24841930
- [Background] Shi E, Shofler D. Maggot debridement therapy: a systematic review. Br J Community Nurs. 2014 Dec;Suppl Wound Care:S6-13. doi: 10.12968/bjcn.2014.19.Sup12.S6. PMID 25478859
- [Background] Sherman RA, Shapiro CE, Yang RM. Maggot therapy for problematic wounds: uncommon and off-label applications. Adv Skin Wound Care. 2007 Nov;20(11):602-10. doi: 10.1097/01.ASW.0000284943.70825.a8. PMID 17975368